CLINICAL TRIAL: NCT03126240
Title: The Role of Sleeve Gastrectomy in Dyslpidemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mohie Eldin, Doctor, Assiut University
Other Study IDs: sleeveindyslipedemia
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sleeve Gastrectomy: This is a five-trocar technique. The abdominal cavity is accessed through a 1cm supraumbilical incision using an optical trocar. The operating ports are inserted under direct vision. The gastroesophageal (GE) junction is exposed. A point on the greater curvature approximately 3-6cm to the pylorus is identified as the distal extent of the resection. Ultrasonic shears are used to divide the vessels long the greater curve up to the angle of His. Linear cutting staplers are used to vertically transect the stomach, creating a narrow gastric tube with. A 19Fr drain is placed in the subhepatic space near the staple line. The resected portion of the stomach is extracted through one of the working ports.

SUMMARY:
The increasing prevalence of obesity noticed in recent decades is a major public health problem of pandemic nature. According to researches, there will be 2.3 billion overweight adults and more than 700 million people suffering from obesity worldwide by the year 2020.Series of epidemiologic studies has revealed a relative link between morbid obesity and metabolic syndrome type 2 diabetes mellitus, hypertension, hyperlipidemia, insulin resistance and shorter life span. Dyslipidemia specially when combined with obesity significantly increase the incidence of atherosclerosis and its complications and also insulin resistance and hence control of diabetic patients. Hyperlipidemia is widely recognized as one of the main co- morbidities in severe obesity and major risk factor for development of atherosclerosis and then heart related diseases.Bariatric surgery has become a prominent treatment modality after the rapidly increasing prevalence of obesity.

DETAILED DESCRIPTION:
The increasing prevalence of obesity noticed in recent decades is a major public health problem of pandemic nature. According to researches, there will be 2.3 billion overweight adults and more than 700 million people suffering from obesity worldwide by the year 2020.Series of epidemiologic studies has revealed a relative link between morbid obesity and metabolic syndrome type 2 diabetes mellitus, hypertension, hyperlipidemia, insulin resistance and shorter life span. Dyslipidemia specially when combined with obesity significantly increase the incidence of atherosclerosis and its complications and also insulin resistance and hence control of diabetic patients. Hyperlipidemia is widely recognized as one of the main co- morbidities in severe obesity and major risk factor for development of atherosclerosis and then heart related diseases[5-6].Bariatric surgery has become a prominent treatment modality after the rapidly increasing prevalence of obesity.

Surgical treatment of higher obesity levels is the most effective procedure due to its simple technique and lower complications with the best outcomes in a long-term perspective. Dramatic weight loss leads to improvement of associated co-morbidities as well. Laparoscopic sleeve gastrectomy leads to long-term weight and improvement or resolution of hypertension, diabetes mellitus type2 and hyperlipidemia.

Studies reported resolution of hypertension in 58% and resolution or improvement of hypertension in 75% of patients following sleeve gastrectomy , resolution of type 2 diabetes mellitus in 84 % of patients as well.

Omana et al. found a greater resolution or improvement of hyperlipidemia with LSG. Hyperlipidemia improved in 87% of patients after LSG.

According to a previous series of studies done before ( 26 studies ) , 11 reported both resolution and improvement of dyslipidemia after LSG and 83.5% of the patients had experienced resolution or improvement of dyslipidemia. Another 7 studies reported only hyperlipidemia resolution and 54% of patients had complete resolution of hyperlipidemia. One study reported improvement of hyperlipidemia in 42% of the patients.

Five studies compared the lipid profile results pre and post-surgery. Only three studies showed minimal changes between pre and post operative cholesterol and LDL levels. However, the same three studies reported significant changes in triglyceride level and HDL level post LSG

ELIGIBILITY:
Inclusion Criteria:

* Have BMI > 40
* Have BMI > 35 with co-morbidities.
* Signed a well informed and signed written consent.
* Patients with abnormal lipid profile
* Patients failed in trials of conservative management including dietary control regarding lipid profile

Exclusion Criteria:

* Endocrine disease
* Severe uncontrolled heart disease
* Inability to follow instruction
* Drug abuse, and cancer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twenty obese patients with an abnormal lipid profile not responding to conservative management will be enrolled in this study
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Low density lipoprotein | at 6 months postoperative
  lipid profile

SECONDARY OUTCOMES:
Low density lipoprotein | at 1 year postoperative
  lipid profile
Total cholesterol level | at 6 months postoperative
  lipid profile
Total cholesterol level | at 1 year postoperative
  lipid profile
High density lipoprotein | at 6 months postoperative
  lipid profile
High density lipoprotein | at 1 year postoperative
  lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohie Eldin, MBBC, Principal Investigator — Specialist

IPD SHARING:
Plan to Share IPD: Undecided